CLINICAL TRIAL: NCT06049381
Title: Tumor Microenvironment Mechanism of LY007 Cell Injection for the Treatment of Relapsed and Refractory B-cell Non-Hodgkin's Lymphoma and the Exploration of Novel CAR-T Translational Research
Brief Title: Tumor Microenvironment Mechanism of LY007 for r/r B-NHL and the Exploration of Novel CAR-T Translational Research
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Principal Investigator, Clinical Professor, Ruijin Hospital
Other Study IDs: LYCAR-01
Record Dates: First submitted 2023-08-28; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Relapsed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients receive LY007 CD20 CAR-T
- Patients receive commerial CD19 CAR-T in China

SUMMARY:
The T cell characteristics of 12 patients treated with CD20 CAR-T (LY007 cell injection) were analyzed to study their relationship with CAR-T anti-tumor activity, tumor killing, and in vivo proliferation, and to explore the mechanisms: before single harvesting, before bridging, before pretreatment, D0, D7, D14, D21, D28, and at the time of follow-up evaluation (plus time points if taking BTKi inhibitors: Peripheral blood specimens were collected before BTKi and 48h after BTKi discontinuation, and peripheral blood cells from patients before and after treatment were analyzed by mass spectrometry flow and single-cell sequencing.

Tumor tissue specimens were collected from patients at different time points (before pretreatment, during CAR-T expansion, and at PD) and subjected to single-cell sequencing.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age (include 18 and 70);
* Eastern Cooperative Oncology Group (ECOG) score of 0-1;
* Cytologically or histologically confirmed diagnosis of CD20-positive B-NHL according to WHO 2016 criteria, including diffuse large B-cell lymphoma (including histologically transformed) and transformed follicular lymphoma (TFL);
* Relapsed or refractory B-cell non-Hodgkin's lymphoma, subjects must have been treated with at least anthracyclines and rituximab (or other CD20-targeted agents) and have relapsed, failed to remit, or progressed after at least second-line therapy or autologous hematopoietic stem cell transplantation (auto-HSCT);

Exclusion Criteria:

* Hepatitis B surface antigen (HBsAg) positive or Hepatitis B core antibody (HBcAb) positive with peripheral blood HBV DNA titer higher than the lower limit of detection; Hepatitis C virus (HCV) antibody positive with HCVRNA titer higher than the lower limit of detection; Human Immunodeficiency Virus (HIV) antibody positive; Positive syphilis serology. 2. Lymphoma involving only the central nervous system (CNS) (subjects with secondary CNS lymphoma are permitted to enroll); and
* Lymphoma involving only the central nervous system (CNS) (subjects with secondary CNS lymphoma are eligible for enrollment). 3. prior CARB vaccination prior to enrollment;
* Prior CAR-T therapy (except for prior targeted CD19 CAR-T therapy, including patients with stable disease evaluated at 3 months after CD19 CAR-T infusion or progressive disease evaluated at any time) or other genetically modified T-cell therapy prior to monotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients from Shanghai Ruijin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression levels of genes (known to be possible driver genes in lymphoma) analyzed from tumor tissues collected before treatment and at the point of progression if available for DNA sequencing after quality control. | 2023.10-2025.12
  Tumor tissues collected before treatment and at the point of progression if available for DNA sequencing after quality control. On the one hand, the difference of tumor mutations will be analyzed in pre-treatment biopsy samples of patients grouped by efficacy; on the other hand, the changes of tumor mutations will be analyzed between pre-treatment and post-treatment biopsy samples of patients.
Expression levels of genes (known to be possible driver genes in lymphoma) analyzed from tumor tissues collected before treatment and at the point of progression if available for RNA sequencing after quality control. | 2023.10-2025.12
  Tumor tissues collected before treatment and at the point of progression if available for bulky RNA sequencing, single-cell RNA sequencing and spatial transcriptome sequencing after quality control. On the one hand, the difference of characteristics of tumor microenvironment will be analyzed in pre-treatment biopsy samples of patients grouped by efficacy; on the other hand, the changes of characteristics of tumor microenvironment will be analyzed between pre-treatment and post-treatment biopsy samples of patients.
Level of M1 macrophage in peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023.10-2025.12
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and immune checkpoints.
Level of M2 macrophage in peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023.10-2025.12
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and immune checkpoints.
Level of OX-40 in peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023.10-2025.12
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and immune checkpoints.
Level of PD-1 in peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023.10-2025.12
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and immune checkpoints.
Level of TIM-3 in peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023.10-2025.12
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and immune checkpoints.
Level of LAG-3 in peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023.10-2025.12
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and immune checkpoints.
Level of lymphocyte subpopulations in peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry. | 2023.10-2025.12
  Peripheral blood collected before each cycle and at the point of progression if available for Mass Cytometry to analyze the changes of immune celltypes and immune checkpoints.

IPD SHARING:
Plan to Share IPD: No